CLINICAL TRIAL: NCT07009574
Title: Factors Associated to Treatment Burden in Patients Affected by Myopic Choroidal Neovascularization
Brief Title: The Treatment Burden of Myopic Choroidal Neovascularization
Acronym: mCNV burden
Status: Not yet recruiting | Type: Observational
Sponsor: Policlinico Gaspare Rodolico - San Marco Catania (Other)
Responsible Party: Principal Investigator, Niccolò Castellino, Assistant Professor of Ophthalmology, Policlinico Gaspare Rodolico - San Marco Catania
Other Study IDs: IRB Catania number 09/2024/PAR
Record Dates: First submitted 2025-05-17; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Myopic Choroidal Neovascularisation; Anti-VEGF Treatment; Burden
Keywords: mcnv; anti-vegf; myopic maculopathy; choroidal neovascularization; myopia
MeSH Terms: conditions — Choroidal Neovascularization; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by myopic choroidal neovascularization
  Interventions: Drug: anti-VEGF intravitreal treatment in patients affected by myopic choroidal neovascularization

INTERVENTIONS:
Drug: anti-VEGF intravitreal treatment in patients affected by myopic choroidal neovascularization — All patients underwent one intravitreal injection at baseline (0.5 mg ranibizumab or 2.0 mg aflibercept); additional intravitreal injections were administered over the follow-up period based on the above-mentioned activity signs with a pro-re-nata (PRN) treatment protocol. The patients have been followed on a monthly or bimonthly basis. The number of visits and examinations in the 12-month study period will be collected.
  Clinical and imaging data of the baseline examination as well as of the 12-month visit (M12) after the first intravitreal injection.

SUMMARY:
Pathologic myopia (PM) is characterized by progressive eye elongation associated with degenerative changes in the retinal and choroidal tissue. Myopic choroidal neovascularization (mCNV) is a well-known complication of PM, occurring in 5-11% of cases and representing a main cause of visual impairment in working people under the age of 50.

The management of patients affected by active mCNV have been revolutionized by the advent of intravitreal injections of anti-vascular endothelial growth factor (anti-VEGF) drugs.

Patients affected by mCNV needs intravitreal injections and visits to assess the need of retreatment with assiduity. It represents a significant burden for patients, caregivers as well as medical equipe.

The aim of this study is to investigate the factors associated with the number of anti-VEGF injections and hospital visits necessary to get mCNV disease stabilization and to identify predictive factors of treatment burden.

DETAILED DESCRIPTION:
Patients affected by treatment-naive mCNV will be included in a 12-month monocentric retrospective cohort study; all patients have been treated with intravitreal anti-VEGF injections between 2020 and 2024 in the Eye Clinic Policlinico Gaspare Rodolico, (Catania, Italy). The study adheres to the tenets of the Helsinki Declaration and ita has been approved by the Institutional review board of the University of Catania (Catania 1 Local Ethical Committee). Informed consent was given by patients at the start of the treatment.

Before starting the treatment, all patients have received a complete ophthalmic examination including a best-corrected visual acuity (BCVA) test, biomicroscopic slit-lamp examination, fundus examination in mydriasis, OCT and OCTA. All patients underwent one intravitreal injection at baseline (0.5 mg ranibizumab or 2.0 mg aflibercept); additional intravitreal injections were administered over the follow-up period according to the activity signs detected (pro-re-nata treatment protocol). Any signs of activity were detected by OCT and OCTA and fluorescein angiography has been performed whenever deemed necessary. Myopic active CNV was defined by clinical (retinal haemorrage detection on fundus examination) and OCT signs (intraretinal cysts, subretinal fluid and subretinal hyperreflective exudation with fuzzy borders). Fluorescein Angiography (FA) was performed .

Clinical and imaging data of the baseline examination and of the 12-month visit (M12) after the first intravitreal injection will be collected.

Best-corrected visual acuity was tested on standard Early Treatment Diabetic Retinopathy Study (ETDRS) charts converted into logarithmic scale of the minimal angle of resolution (logMAR). OCT and FA were carried out by Spectralis HRA+OCT with a confocal scanning laser ophthalmoscope (Heidelberg Engineering, Heidelberg, Germany). The OCT scan protocol used was a 15°x15° 67-section macular cube with additional high resolution horizontal and vertical single lines centred on the CNV. AngioVue XR Avanti (Optovue Inc, Fremont, California, USA) was employed to perform OCTA. A light source of 840 nm was used and the A-scan rate was 70,000 per second with a bandwidth of 50 nm. The macula images (6mmx6mm) obtained by OCTA were centered on the foveola. Each volume contained 400x400 A-scans with two consecutive B-scans acquired in each fixed position. The split-spectrum amplitude-decorrelation angiography (SSADA) method was used to capture the dynamic motion of red blood cells. mCNV areas were selected manually using AngioAnalytics software on the outer retina slab.

The values of the "CNV select area" will be included in the analysis as mCNV size. The Central Macular Thickness (CMT, micron) automatically provided by the machine, will be collected.

Myopic CNV will be categorized either as subfoveal (the CNV reaches the center of the fovea) or juxtafoveal (less than 200 micron from the center of the fovea) according to the location. In addition, mCNV will be categorized by OCTA features, either as immature (small-size, poorly structured neovascular network), or mature (larger and fully organized neovascular network) according to previous findings. Subretinal fibrosis (SF) will be defined as the detection at fundus examination of yellowish or greyish subretinal tissue in the foveal or parafoveal area, corresponding to an OCT image of a well-demarcated hyperreflective lesion situated between the retinal pigment epithelium and the neurosensory retina.

The number of in-hospital visits, invasive imaging examination (fluorescein angiography) as well as the number of intravitreal injections that underwent the patient will be collected and represent the burden of treatment.

The following clinical and imaging parameters will be included in the analysis: sex, age (years), anti-VEGF drug administered, mCNV location (subfoveal or juxtafoveal). BCVA (logMAR), CNV area (mm2), mCNV pattern will be assessed both at baseline visit and at 12-month visit. At the end of the follow-up period (12 months) will be assessed the presence of subretinal fibrosis (SF). The eyes will be categorized as stable (number of injections ≤ 2) or unstable (number of injections > 2) according to the number of injections administered as previously reported).

All the data will be collected according to the above-mentioned criteria by using a standardized Excel spreadsheet (Microsoft Corp.). In case of lacking data the patient will be excluded from the study.

Statistical analysis will be performed by SPSS (version 22, IBM, New York, USA). Variables related to the number of injections at 12 months (dependent variable) will be tested in a univariate regression analysis; any variable with a p value <0.2 in univariate analysis will be included in multivariate logistic regression analysis. Comparison of continuous variable values between two groups will be performed by unpaired t-test. Potential risk factors for more than 2 injections (unstable group) will be identified in univariate analyses, using the chi-square or Fisher exact tests for categorical variables, and Mann-Whitney tests for quantitative variables. Odd ratio will be calculated, and Exp(B) from binary logistic regression will be used for the continuous variables. P-values lower than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* axial length>26 mm or refractive error (spherical equivalent) <-6 Diopters
* clinical changes typical of Pathologic myopia
* diagnosis of subfoveal or juxtafoveal treatment-naïve myopic choroidal neovascularization (mCNV)
* only one eye per patient was included in the analysis, in cases of patients treated bilaterally only the first eye treated was included

Exclusion Criteria:

* Extrafoveal mCNV location
* Other retinal diseases
* any inflammatory condition which may cause CNV including multifocal choroiditis, puntate inner choroidopathy and white dot syndrome
* previous ocular surgery (except for cataract extraction performed before the baseline visit)
* inferior quality imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by myopic choroidal neovascularization
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
To assess treatment burden | one year
  The number of access of the patient to the hospital for any clinical need (intravitreal injections administration, imaging examinations and visits) in the first year of anti-VEGF treatment.

SECONDARY OUTCOMES:
Visual Acuity | one year
  Visual acuity (logMAR)
Intraretinal Cysts | one year
  Presence of intraretinal cysts detected by OCT
Subretinal fluid | one year
  Presence of OCT subretinal fluid by OCT
Subretinal fuzzy material | one year
  Presence of subretinal fuzzy material detected by OCT
Subretinal fibrosis | one year
  Presence of subretinal fibrosis betected by OCT
Cnv maturity pattern | one year
  Assessment of the maturity pattern of the myopic choroidal neovascularization detected by OCT (Mature/Immature)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Rodolico, Catania, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided